CLINICAL TRIAL: NCT06143436
Title: A Study on the Correlation Between TCM Constitution, Pattern Types, and Disease Factors in Primary Lung Cancer.
Brief Title: TCM Constitution, Pattern Types, and Disease Factors in Primary Lung Cancer.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH112-REC3-157
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Medicine, Chinese Traditional; Body Constitution; Syndrome; Risk Factors
MeSH Terms: conditions — Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Constitution in Chinese Medicine Questionnaire — Using questionnaire to collect data from new lung cancer patients.

SUMMARY:
Recently, TCM has played an important role in adjuvant therapy for lung cancer. TCM treatment is based on pattern identification, and constitution theory is also used as a tool for TCM to predict the disease progression. Although there have been many researchs related to the pattern identification and constitution of lung cancer, in view of the problems and limitations, further research on lung cancer patients in Taiwan is needed.

This study aims to explore the correlation between TCM constitution, pattern identification, and other related factors in patients with primary lung cancer in Taiwan, hoping to reveal the disease characteristics of lung cancer in TCM theory. This study intends to interview subjects through attending physicians in the thoracic ward and outpatient clinic of the CMUH from November 20th, 2023 to May 19th , 2025, and the subjects will be included in this study after the researchers ask the subjects for consent.

This study will collect the demographic data of the subjects (sex, age, BMI, smoking history) and disease-related clinical data (tumor stage, pathological type, gene mutation, tumor markers, other comorbidities), and the investigator will ask about the subjects' signs according to the Constitution in Chinese Medicine Questionnaire (CCMQ) , ask the subjects' symptoms according to the pattern identification table, obtain the data to analyze their distribution by descriptive statistics, and then analyze the correlation between them by analysis of variance and Chi-square test.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with primary lung cancer.
* Age greater than 18 years and less than 100 years.
* After explanation, they agree to join this study and voluntarily sign the subject consent form, and can understand the content of the questionnaire.

Exclusion Criteria:

* Pregnant women.
* Severe mental illness that affects the response to the questionnaire.
* Has been treated (e.g., surgery, chemotherapy, targeted therapy, immunotherapy, radiation therapy, etc.).
* Concomitant with other uncured primary malignancies.
* Patients with other serious primary diseases (such as: liver and kidney dysfunction, hematolymphatic system diseases, etc.).
* Severe respiratory diseases that are not lung cancer (e.g. primary emphysema, interstitial fibrosis, etc.) .

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with primary lung cancer without any treatment.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2025-05-19 (Estimated); Study Completion 2025-05-19 (Estimated)

PRIMARY OUTCOMES:
TCM body constitution | 20-30 minuts
  Ask about the subjects' signs according to the Constitution in Chinese Medicine Questionnaire (CCMQ)
TCM pattern types | 20-30 minuts
  Ask about the subjects' symptoms according to the pattern identification table

SECONDARY OUTCOMES:
demographic data | 1 day
  sex, age, BMI, smoking history
disease-related clinical data | 1 day
  tumor stage, pathological type, gene mutation, tumor markers, other comorbidities

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan